CLINICAL TRIAL: NCT02221336
Title: Daily Electronic Monitoring of Subjective and Objective Measures of Illness Activity in Bipolar Disorder - The MONARCA II Trial (MONitoring, treAtment and pRediCtion of bipolAr Disorder Episodes II)
Brief Title: Daily Subjective and Objective Smartphone Measures of Illness Activity to Treat Bipolar Disorder- The MONARCA II Trial
Acronym: MONARCAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: University of Copenhagen (Other); IT University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Faurholt-Jepsen, Principal Investigator, MD and PhD student, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2014-059
Record Dates: First submitted 2014-08-12; First posted 2014-08-20 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Daily electronic monitoring; Smartphones; Subjective and objective smartphone data; Feedback loop
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-MONARCA II system (Placebo Comparator): Use of smartphone for normal communicative purposes only. No self-monitoring and no feedback loop.
  Interventions: Device: Non-MONARCA II system
- The MONARCA II system (Experimental): Daily electronic monitoring of subjective and objective smartphone measures including a feedback loop
  Interventions: Device: The MONARCA II system

INTERVENTIONS:
Device: The MONARCA II system — Daily electronic monitoring of subjective and objective smartphone measures including a feedback loop
  Other Names: Non-MONARCA II system (control group condition)
  Arms: The MONARCA II system
Device: Non-MONARCA II system — Daily use of smartphone for normal communicative purposes. No self-monitoring in the MONARCA II system.
  Arms: Non-MONARCA II system

SUMMARY:
Bipolar disorder is associated with a high risk of relapse and hospitalisation and many patients do not recover to their previous psychosocial function. Major reasons for poor outcomes are delayed intervention for prodromal depressive and manic symptoms as well as decreased adherence with treatment.

Recently, in the MONARCA I trial (NCT01446406), the investigators developed and deployed a smartphone based self-monitoring system (the MONARCA I system) in a randomized controlled trial, to test the effect of daily reporting of subjective self-monitoring of depressive and manic symptoms as well as a bi-directional feedback loop on depressive and manic symptoms.

In the MONARCA II trial the investigators will develop and deploy a new version of the smartphone based monitoring system. The investigators will in a randomized controlled single blind trial investigate whether daily electronic monitoring of subjective and objective measures of illness activity using a smartphone based self-monitoring system including feedback on subjective as well as automatically generated objective data (e.g.social activity, physical activity etc.) (the MONARCA II system) reduces the severity of depressive and manic symptoms and improves functioning more than a control group receiving a smartphone. All patients will be followed for 9 months with outcome assessments at baseline, after 4 weeks, after 3 months, after 6 months and after 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Disorder according to SCAN interview
* ≥18 years of age
* Patients who previously have received a course of treatment at the Clinic for Affective Disorders, Psychiatric Centre Copenhagen, Denmark

Exclusion Criteria:

* Pregnancy
* Lack of Danish language skills
* Patients who previously have received and used the MONARCA I system for self-monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Differences between the groups in depressive and manic symptoms and the number of affective episodes | Baseline and up to 9 months
  Differences between the groups in depressive and manic symptoms measured using Hamilton Depression Rating Scale (HDRS) and Young Mania Rating Scale (YMRS) and episodes defined ad HDRS<= 14 and/or YMRS<= 14

SECONDARY OUTCOMES:
Differences between the groups in smartphone measures | Baseline and up to 9 months
  Differences between the groups in:
  -Automatically generated objective smartphone measures
Differences between the groups in number of hospitalizations | Baseline up to 9 months follow up
  Differences between the groups in number of hospitalization
Differences between the groups in number of contacts to clinicians and emergency rooms | Baseline up to 9 months follow up
  Differences between the groups in number of contacts to clinicians and emergency rooms
Differences between the groups in functioning | Baseline up to 9 months follow up
  Differences between the groups in functioning measured using the FAST questionnaire
Differences between the groups in perceived stress | Baseline up to 9 months
  Differences between the groups in perceived stress using the perceived stress questionnaire
Differences between the groups in quality of life | Baseline up to 9 months follow up
  Differences between the groups in quality of life measured using the WHOQoL questionnaire
Differences between the groups in self-rated depressive symptoms | Baseline up to 9 months
  Differences between the groups in self-rated depresisve symptoms using the BDI questionnaire
Differences in self-rated manic symptoms | Baseline up to 9 months follow up
  Differences between the groups in self-rated manic symptoms using the ASRM questionnaire
Differences between the groups in adherence to medication | Baseline up to 9 months follow up
  Differences between the groups in adherence to medication measured using the questionnaire MARS
Differences between the groups in recovery | Baseline up to 9 months follow up
  Differences between the groups in recovery using the questionnaire Recovery Assessment Scale (RAS)
Differences between the groups in empowerment | baseline up ot 9 months
  Differences between the groups in empowerment using the questionnaire Rogers Empowerment scale.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Faurholt-Jepsen, MD, Principal Investigator — Psychiatric Centre Copenhagen, Rigshospitalet, Denmark
Locations (1):
- Psychiatric Centre Copenhagen, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Faurholt-Jepsen M, Frost M, Vinberg M, Christensen EM, Bardram JE, Kessing LV. Smartphone data as objective measures of bipolar disorder symptoms. Psychiatry Res. 2014 Jun 30;217(1-2):124-7. doi: 10.1016/j.psychres.2014.03.009. Epub 2014 Mar 13. PMID 24679993
- [Background] Faurholt-Jepsen M, Vinberg M, Christensen EM, Frost M, Bardram J, Kessing LV. Daily electronic self-monitoring of subjective and objective symptoms in bipolar disorder--the MONARCA trial protocol (MONitoring, treAtment and pRediCtion of bipolAr disorder episodes): a randomised controlled single-blind trial. BMJ Open. 2013 Jul 24;3(7):e003353. doi: 10.1136/bmjopen-2013-003353. Print 2013. PMID 23883891
- [Derived] Faurholt-Jepsen M, Frost M, Christensen EM, Bardram JE, Vinberg M, Kessing LV. Validity and characteristics of patient-evaluated adherence to medication via smartphones in patients with bipolar disorder: exploratory reanalyses on pooled data from the MONARCA I and II trials. Evid Based Ment Health. 2020 Feb;23(1):2-7. doi: 10.1136/ebmental-2019-300106. PMID 32046986
- [Derived] Faurholt-Jepsen M, Frost M, Busk J, Christensen EM, Bardram JE, Vinberg M, Kessing LV. Differences in mood instability in patients with bipolar disorder type I and II: a smartphone-based study. Int J Bipolar Disord. 2019 Feb 1;7(1):5. doi: 10.1186/s40345-019-0141-4. PMID 30706154
- [Derived] Faurholt-Jepsen M, Vinberg M, Frost M, Christensen EM, Bardram J, Kessing LV. Daily electronic monitoring of subjective and objective measures of illness activity in bipolar disorder using smartphones--the MONARCA II trial protocol: a randomized controlled single-blind parallel-group trial. BMC Psychiatry. 2014 Nov 25;14:309. doi: 10.1186/s12888-014-0309-5. PMID 25420431